CLINICAL TRIAL: NCT04264234
Title: Management Of Placenta Previa Cases And Determination Of Hospitalization Criteria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Sabahattin Anıl Arı, Principal Investigator, Ege University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-9.1/27
Record Dates: First submitted 2018-11-03; First posted 2020-02-11 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Placenta Previa
Keywords: placenta previa; placental invasion anomalies; timing of the birth
MeSH Terms: conditions — Placenta Previa | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: Placenta previa cases will be followed up at 28th gestational week and evaluated at 32nd week by vaginal ultrasonography and MRI and this follow-up will continue until delivery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Placenta Previa (Experimental): Placenta previa cases will be evaluated at 32nd week by vaginal ultrasonography and MRI.
  Interventions: Diagnostic Test: Vaginal Ultrasonography; Diagnostic Test: Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Vaginal Ultrasonography — Placenta previa cases will be evaluated at 32nd week by vaginal ultrasonography for invasion anomaly and preterm birth.
Diagnostic Test: Magnetic Resonance Imaging — Placenta previa cases will be evaluated at 32nd week by MRI for invasion anomaly and preterm birth.

SUMMARY:
Placenta previa cases are one of the difficult groups of patients to manage in modern obstetrics. When the literature is evaluated extensively, no clear information can be seen especially in terms of hospitalization time. Inpatient follow-up of this patients has negative effects like hospital infections in terms of the patient, workload in terms of health personnel and financial losses in terms of the country's economy. Placenta previa cases are complicated patients in which generalizations cannot be easily performed and they should be monitored at third level hospitals. In addition, care should be personalized considering the many reasons. In this study, placenta previa cases will be followed up at 28th gestational week and evaluated at 32nd week by vaginal ultrasonography and MRI and this follow-up will continue until delivery. Thus, in this study, it was aimed to determine the parameters that would allow systematic personalization of health service in this particular patient group by making risk assessment of placenta previa cases.

ELIGIBILITY:
Inclusion Criteria:

* Monitoring of placenta previa
* To apply before the 28th week
* To have a low-risk second trimester screening test
* No malformation detected in the anomaly screening

Exclusion Criteria:

* Multiple pregnancies
* Pregnancy complicated with preeclampsia
* Pregnancy complicated by gestational hypertension
* Pregnancy complicated by gestational diabetes mellitus

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant participant
Enrollment: 98 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
The number of placental invasion pathologies | 1 day
  Placental invasion pathologies detected during delivery will be evaluated.
The number of preterm birth | 1 day
  The relation between preterm birth and placental invasion pathologies will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Sabahattin a Arı, MD, Principal Investigator — Ege University
Locations (1):
- Ege University Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No